CLINICAL TRIAL: NCT05849441
Title: Online Mindfulness Intervention for Adolescents With 22q11DS
Brief Title: Mindfulness Program for Adolescents With 22q11DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MindfulnessinTeens-SBIR-23-001
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: 22Q11 Deletion Syndrome
MeSH Terms: conditions — 22q11 Deletion Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online mindfulness intervention (Experimental): Participants will have access to the intervention between pre-test and post-test assessments. The intervention, Aware Program, is an online mindfulness education program for adolescents with 22q11DS designed to enhance their coping skills and ability to manage stress and anxiety in healthy ways.
  Interventions: Behavioral: Aware Program
- Wait-List Control (No Intervention): Participants will not have access to the online mindfulness intervention between the pre-test and post-test assessments. After completing the post-test questionnaires, participants in the wait-list control group will receive access to the online mindfulness intervention (Aware Program).

INTERVENTIONS:
Behavioral: Aware Program — The program includes interactive, multimedia lessons for adolescent participants to learn, practice, and apply different mindfulness skills. Parent-adolescent pairs will have the option to subscribe to a mobile messaging service that includes progress reminders, encouragement, and practice content. Parent participants also have access to online resources to support and monitor their teen's use of the program.
  Arms: Online mindfulness intervention

SUMMARY:
The goal of this study is to evaluate the effectiveness of the Aware Program, an online mindfulness education program, with adolescents with 22q11DS and their parents.

DETAILED DESCRIPTION:
Parent-adolescent pairs (N=60) will be recruited to participate in a randomized controlled trial. Consent, permission, and/or assent will be sought prior to participation in the study. Participant pairs will be randomized into one of two study arms: intervention and wait-list control. All participants will complete a web-based pre-test questionnaire. Adolescents and parents in the intervention group will then receive access to the Aware Program for four weeks. Approximately 4-5 weeks after completing the pre-test questionnaire, all participants will complete a web-based post-test questionnaire (the post-test for the intervention group will include Consumer Satisfaction questions about the program). Adolescents and parents in the wait-list control group will then have the option of reviewing the Aware Program and will receive access for four weeks. After approximately four weeks, they will have the opportunity to complete the Consumer Satisfaction Questionnaire about the program.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, youth must:

* Have received a diagnosis of 22Q11.DS (also known as VeloCardioFacial Syndrome or DiGeorge syndrome)
* Be between the ages of 12 and 19 years old
* Have an IQ of greater than or equal to 55
* Have regular internet and computer access
* Speak and read English (all study and program materials are in English)

To be included in the study, parents must:

* Have a participating youth in the study
* Read fluently in English (all study and program materials are in English)

Exclusion Criteria:

- Only one parent per youth may participate

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Parker, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 parent-adolescent pairs (which totals 110 participants) were randomized to condition (intervention or wait-list control).
Period: Overall Study
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Started | 54 (27 adolescents and 27 parents) | 56 (28 adolescents and 28 parents)
Completed Pretest | 50 (25 adolescents and 25 parents) | 54 (27 adolescents and 27 parents)
Completed | 42 (21 adolescents and 21 parents) | 54 (27 adolescents and 27 parents)
Not Completed | 12 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Mindfulness Intervention | Wait-List Control | Total
Number analyzed (Participants) | 50 | 54 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall sample includes parents and adolescents. The analysis population for adolescent age includes just adolescents and the analysis population for parent age includes just parents.
  years
    Adolescent: number analyzed (Participants) | 25 | 27 | 52
    Adolescent | 14.52 (2.18) | 14.92 (1.75) | 14.73 (1.96)
    Parent: number analyzed (Participants) | 25 | 27 | 52
    Parent | 46.04 (8.02) | 51.30 (8.00) | 48.77 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. The adolescent sex/gender categories only include adolescents and the parent sex/gender categories only include parents.
  Participants
    Adolescent: number analyzed (Participants) | 25 | 27 | 52
    Adolescent: Female | 13 | 10 | 23
    Adolescent: Male | 12 | 17 | 29
    Parent: number analyzed (Participants) | 25 | 27 | 52
    Parent: Female | 24 | 26 | 50
    Parent: Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. The adolescent ethnicity categories include only adolescents and the parent ethnicity categories include only parents.
  Participants
    Adolescent: number analyzed (Participants) | 25 | 27 | 52
    Adolescent: Hispanic or Latino | 5 | 0 | 5
    Adolescent: Not Hispanic or Latino | 19 | 26 | 45
    Adolescent: Unknown or Not Reported | 1 | 1 | 2
    Parent: number analyzed (Participants) | 25 | 27 | 52
    Parent: Hispanic or Latino | 1 | 1 | 2
    Parent: Not Hispanic or Latino | 24 | 26 | 50
    Parent: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. The adolescent race categories include only adolescents and the parent race categories include only parents.
  Participants
    Adolescent: number analyzed (Participants) | 25 | 27 | 52
    Adolescent: American Indian or Alaska Native | 1 | 1 | 2
    Adolescent: Asian | 2 | 3 | 5
    Adolescent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescent: Black or African American | 2 | 1 | 3
    Adolescent: White | 19 | 19 | 38
    Adolescent: More than one race | 1 | 1 | 2
    Adolescent: Unknown or Not Reported | 0 | 2 | 2
    Parent: number analyzed (Participants) | 25 | 27 | 52
    Parent: American Indian or Alaska Native | 0 | 0 | 0
    Parent: Asian | 2 | 2 | 4
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 0 | 1 | 1
    Parent: White | 21 | 22 | 43
    Parent: More than one race | 2 | 2 | 4
    Parent: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 54 | 104
Adolescent psychological diagnosis [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. This item only asked about the adolescents' psychological diagnosis.
  Participants
    number analyzed (Participants) | 25 | 27 | 52
    Yes | 20 | 20 | 40
    No | 5 | 7 | 12
Parent education [Count of Participants; unit: Participants] — Population: The overall sample includes parents and adolescents. This item only asked about the parents' education.
  Participants
    number analyzed (Participants) | 25 | 27 | 52
    No college degree or less | 10 | 4 | 14
    College degree or higher | 15 | 23 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adolescents' Coping Skills
Description: Adolescents will be asked to respond to 34 questions (e.g., Try to think of different ways to solve it; 1 = Never; 5 = Always) that assess their coping in response to stressors across 5 domains: Seeking Social Support, Problem Solving, Distancing, Externalizing, and Internalizing. Three items related to mindfulness skills will be included as a mindfulness subscale. Responses will be averaged across each domain and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater use of the coping strategy.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale
  Support Seeking | 3.10 (.15) | 2.68 (.13)
  Problem Solving | 3.18 (.12) | 2.79 (.11)
  Distancing | 2.67 (.09) | 2.60 (.08)
  Internalizing | 2.69 (.11) | 2.64 (.10)
  Externalizing | 2.41 (.12) | 2.42 (.11)
  Mindfulness | 3.11 (.16) | 2.73 (.15)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.04, Regression, Linear — This is for the subscale: Support-Seeking
Statistical Analysis 2: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.02, Regression, Linear — This is for subscale: Problem Solving
Statistical Analysis 3: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.55, Regression, Linear — This is for subscale: Distancing
Statistical Analysis 4: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.79, Regression, Linear — This is for subscale: Internalizing
Statistical Analysis 5: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.93, Regression, Linear — This is for subscale: Externalizing
Statistical Analysis 6: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.09, Regression, Linear — This is for subscale: Mindfulness

2. Primary Outcome: Change From Baseline in Adolescents' Emotion Regulation
Description: Adolescents will be asked to respond to 10 questions (e.g., I keep my emotions to myself; 1 = Strongly disagree; 7 = Strongly agree) that assess their use of two emotion regulation strategies: Cognitive Reappraisal and Suppression. Responses will be averaged across each strategy and the minimum scale is 1 and the maximum scale score is 7. Higher scores indicate greater use of the emotion regulation strategy.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale
  Reappraisal | 4.49 (.21) | 4.21 (.18)
  Suppression | 3.59 (.19) | 3.28 (.17)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.32, Regression, Linear — This is for subscale: Reappraisal
Statistical Analysis 2: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.24, Regression, Linear — This is for subscale: Suppression

3. Primary Outcome: Change From Baseline in Adolescents' Emotional Self-efficacy
Description: Adolescents will be asked to respond to 27 questions (e.g., I can tell when my feelings change; 1 = Not confident at all; 5 = Very confident) that assess their beliefs about their ability to understand and manage emotions. The measure has four factors: Using and managing your own emotions; Identifying and understanding your own emotions; Dealing with emotions in others; Perceiving emotion through facial expressions and body language. Responses will be averaged across the four factors and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater emotional self-efficacy.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale
  Manage own emotions | 3.33 (.10) | 3.24 (.09)
  Identify and understand own emotions | 3.70 (.14) | 3.96 (.12)
  Deal with emotions of others | 3.21 (.11) | 3.38 (.10)
  Perceive emotion through faces and bodies | 3.40 (.16) | 3.51 (.14)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.53, Regression, Linear — This is for subscale: Manage own emotions
Statistical Analysis 2: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.16, Regression, Linear — This is for subscale: Identify and Understand Own Emotions
Statistical Analysis 3: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.27, Regression, Linear — This is for subscale: Deal with emotions of others
Statistical Analysis 4: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.59, Regression, Linear — This is for subscale: Perceive emotions through faces and bodies

4. Primary Outcome: Change From Baseline in Adolescents' General Anxiety
Description: Adolescents will be asked to respond to 7 items that assess general anxiety (e.g., Over the last two weeks, how often have you been bothered by the following problems… feeling nervous, anxious, or on edge; 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day). Responses will be summed across the 7 items and the minimum scale score is 0 and the maximum scale score is 21. Higher scores indicate greater general anxiety.
Time Frame: Baseline and Week 4
Population: Missing data from two adolescents
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 20 | 26
units on a scale | 5.90 (1.07) | 8.08 (.92)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.16, Regression, Linear

5. Primary Outcome: Change From Baseline in Adolescents' Social Anxiety
Description: Adolescents will be asked to respond to 18 items (e.g., It's hard for me to ask others to do things with me; 1 = Not at all; 5 = All the time) that assess social anxiety. The measure has three factors: Fear of Negative Evaluation, Social Avoidance and Distress-New; Social Avoidance and Distress. Responses will be summed across each of the three factors. The minimum scale score is 1 and the maximum scale score is 40. Higher scores indicate greater social anxiety.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale
  Fear of negative evaluation | 23.06 (1.49) | 22.14 (1.32)
  Social avoidance and distress (new) | 19.68 (1.06) | 20.43 (.94)
  Social avoidance and distress (general) | 11.62 (.65) | 10.56 (.57)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.65, Regression, Linear — This is for subscale: Fear of Negative Evaluation
Statistical Analysis 2: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.60, Regression, Linear — This is for subscale: Social avoidance and distress (new)
Statistical Analysis 3: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.23, Regression, Linear — This is for subscale: social avoidance and distress (general)

6. Primary Outcome: Change From Baseline in Adolescents' Wellbeing
Description: Adolescents will be asked to respond to a total of 7 items that assess their overall health and wellbeing using the PROMIS Pediatric Scale - Global Health 7 measure. Adolescents will respond to 4 items (e.g., In general, would you say your quality of life is…; 5 = Excellent, 1 = Poor); 1 item (e.g., How often do you feel really sad; 5 = Never; 1 = Always); and 2 items (e.g., How often do you have fun with friends?; 5 = Always; 1 = Never). Responses were summed across the 7 items to create a single global health score. The scoring table in the PROMIS Global Health Scoring manual was used to convert a summed global health score into a T score value for each participant. The T score has a mean of 50 with a standard deviation of 10. Higher T scores on this measure represent greater adolescent overall health and wellbeing.
Time Frame: Baseline and Week 4
Population: All 7 items in this measure had to be answered in order to produce a valid global health T score. If a participant did not answer all 7 questions, no score was included in the dataset. Thus, 4 participants were excluded from the analysis of this measure.
Measure: Least Squares Mean (Standard Error); unit: T score
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 19 | 25
T score | 45.60 (1.86) | 47.11 (1.62)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.55, Regression, Linear

7. Primary Outcome: Change From Baseline in Parent Report of Adolescents' Emotion Regulation
Description: Parents will be asked to respond to 24 questions (e.g., Responds positively to neutral or friendly overtures by peers; 1= Never; 4 = Always) that assess parent ratings of their adolescents' emotion regulatory abilities. There are two subscales for this measure: Emotion Regulation and Negativity. Responses will be averaged across the two subscales and the minimum scale score is 1 and the maximum scale score is 4. Higher scores indicate greater use of the emotion regulation strategy.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale
  Negativity | 2.05 (.05) | 2.17 (.05)
  Emotion Regulation | 2.82 (.06) | 2.84 (.05)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.11, Regression, Linear — This is for subscale: Negativity
Statistical Analysis 2: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.79, Regression, Linear — This is for subscale: Emotion regulation

8. Primary Outcome: Change From Baseline in Parent Report of Adolescents' Executive Functioning
Description: Parents will be asked to respond to 24 questions (e.g., Has difficulty thinking ahead or learning from experience; 1 = Definitely not true; 5 = Definitely true) that assess parent ratings of their adolescents' executive functioning. There are four subscales: Working Memory, Planning, Inhibition, and Regulation. Responses will be averaged across the four subscales and the minimum scale score is 1 and the maximum scale score is 5. Higher scores indicate greater executive functioning deficit.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale
  Working Memory | 3.54 (.10) | 3.73 (.08)
  Planning | 3.71 (.13) | 3.93 (.12)
  Inhibit | 2.96 (.09) | 3.04 (.08)
  Regulate | 3.93 (.13) | 4.09 (.11)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.14, Regression, Linear — This is for subscale: Working Memory
Statistical Analysis 2: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.20, Regression, Linear — This is for subscale: Planning
Statistical Analysis 3: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.48, Regression, Linear — This is for subscale: Inhibit
Statistical Analysis 4: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.37, Regression, Linear — This is for subscale: Regulation

9. Primary Outcome: Change From Baseline in Parent Report of Adolescents' Anxiety
Description: Parents will be asked to respond to 8 questions (e.g., My child worries about things; 0 = Never; 3 = Always) that assess parent ratings of their adolescents' anxiety. Responses will be summed across the 8 items and the minimum scale score is 0 and the maximum scale score is 24. Higher scores indicate greater anxiety.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
units on a scale | 8.59 (.48) | 8.10 (.42)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.45, Regression, Linear

10. Primary Outcome: Change From Baseline in Parent Report of Adolescents' Wellbeing
Description: Parents will be asked to respond to a total of 7 items that assess parent ratings of their adolescents' overall health and wellbeing using the PROMIS Parent Proxy Scale - Global Health 7. Parents will respond to 4 items (e.g., In general, would you say your child's quality of life is…; 5 = Excellent, 1 = Poor); 1 item (e.g., How often does your child feel really sad; 5 = Never; 1 = Always); and 2 items (e.g., How often does your child have fun with friends?; 5 = Always; 1 = Never). Responses were summed across the 7 items to create a single global health score. The scoring table in the PROMIS Global Health Scoring manual was used to convert a summed global health score into a T score value for each participant. The T score has a mean of 50 with a standard deviation of 10. Higher T scores on this measure represent greater adolescent overall health wellbeing as rated by their parent.
Time Frame: Baseline and Week 4
Measure: Least Squares Mean (Standard Error); unit: T score
Arm/Group | Online Mindfulness Intervention | Wait-List Control
Number analyzed (Participants) | 21 | 27
T score | 37.88 (.82) | 37.71 (.73)
Statistical Analysis 1: Comparison: Online Mindfulness Intervention vs Wait-List Control; Test type: Superiority; p = 0.88, Regression, Linear

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The participants in the study completed web-based questionnaires and utilized an online mindfulness education program (if in the intervention group). The risks associated with this study were minimal and the participants were not at risk for mortality as a function of participating in this study. Because this study investigated an online behavioral intervention, All-Cause Mortality was not monitored or assessed.
Arm/Group | Online Mindfulness Intervention | Wait-List Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/54
Other Adverse Events (participants affected / at risk) | 0/50 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT05849441/Prot_SAP_000.pdf